CLINICAL TRIAL: NCT01674647
Title: A Prospective, Randomized, Open-label, Parallel-group, Active-controlled, Multicenter Study Exploring the Efficacy and Safety of Once-daily Oral Rivaroxaban (BAY59-7939) Compared With That of Dose-adjusted Oral Vitamin K Antagonists (VKA) for the Prevention of Cardiovascular Events in Subjects With Nonvalvular Atrial Fibrillation Scheduled for Cardioversion
Brief Title: Explore the Efficacy and Safety of Once-daily Oral Rivaroxaban for the Prevention of Cardiovascular Events in Subjects With Nonvalvular Atrial Fibrillation Scheduled for Cardioversion
Acronym: X-VERT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15693; 2011-002234-39 (EudraCT Number)
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Results first posted 2015-02-03 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Atrial Fibrillation
Keywords: rivaroxaban; oral anticoagulant; nonvalvular atrial fibrillation; cardioversion; stroke; transient ischemic attack; thromboembolism; cardiovascular event
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Ischemic Attack, Transient; Thromboembolism | interventions — Rivaroxaban; acarboxyprothrombin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Xarelto, BAY59-7939) (Experimental): A Direct Cardioversion Strategy can be performed only if sufficient anticoagulation is proven during the last 21 days prior to randomization and/or a transesophageal echocardiogram (TEE) is planned before cardioversion. Rivaroxaban will be given for 1-5 days before planned direct cardioversion. The run-in of 1-5 days is needed due to potential pretreatment with VKA. Treatment with rivaroxaban will be continued for 42 days after the cardioversion. A Delayed Cardioversion Strategy will be chosen if sufficient anticoagulation is not proven during the last 21 days prior to randomization and no TEE is planned. Rivaroxaban will be given for at least 21 (+4) days before the planned cardioversion, to a maximum of 56 (+4) days prior to planned cardioversion.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Vitamin K antagonist (VKA) (Active Comparator): A Direct Cardioversion Strategy can be performed only if sufficient anticoagulation is proven during the last 21 days prior to randomization and/or a transesophageal echocardiogram (TEE) is planned before cardioversion. VKA will be given for 1-5 days before planned direct cardioversion. The run-in of 1-5 days is needed due to potential pretreatment with VKA. Treatment with VKA will be continued for 42 days after the cardioversion. A Delayed Cardioversion Strategy will be chosen if sufficient anticoagulation is not proven during the last 21 days prior to randomization and no TEE is planned. VKA will be given for at least 21 (+4) days before the planned cardioversion, to a maximum of 56 (+4) days prior to planned cardioversion.
  Interventions: Drug: Vitamin K antagonist (VKA)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Rivaroxaban 20 mg orally once daily; subjects with moderate renal impairment (ie, CrCl of 30 to 49 mL/min, inclusive) will receive the adjusted dose of 15 mg orally once daily in the study
  Arms: Rivaroxaban (Xarelto, BAY59-7939)
Drug: Vitamin K antagonist (VKA) — VKA orally once daily titrated to a target international normalized ratio (INR) of 2.5 (range 2.0-3.0, inclusive); the VKA type (eg, warfarin, acenocoumarol, phenprocoumon, fluindione, etc) will be assigned by the investigator according to local treatment standards
  Arms: Vitamin K antagonist (VKA)

SUMMARY:
A study for patients with abnormal heart rhythm (atrial fibrillation) who need to undergo cardioversion (procedure to restore normal heart rhythm). The study will compare patients assigned randomly (like flipping a coin) to either Rivaroxaban or vitamin K antagonist (VKA). The study will measure common medical outcomes for this type of patient such as bleeding and stroke.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged >= 18 years
* Hemodynamically stable nonvalvular atrial fibrillation longer than 48 hours or of unknown duration
* Scheduled for cardioversion (electrical or pharmacological) of nonvalvular atrial fibrillation
* Women of childbearing potential and men must agree to use adequate contraception when sexually active

Exclusion Criteria:

* Severe, disabling stroke (modified Rankin score of 4- 5, inclusive) within 3 months or any stroke within 14 days prior to randomization
* Transient ischemic attack within 3 days prior to randomization
* Acute thromboembolic events or thrombosis (venous/arterial) within the last 14 days prior to randomization
* Acute Myocardial infarction (MI) within the last 14 days prior to randomization
* Cardiac-related criteria: known presence of cardiac thombus or myxoma or valvular atrial fibrillation
* Active bleeding or high risk for bleeding contraindicating anticoagulant therapy
* Concomitant medications: indication for anticoagulant therapy other than atrial fibrillation, chronic aspirin therapy > 100 mg daily or dual antiplatelet therapy, strong inhibitors of both cytochrome P450 (CYP) 3A4 and P-glycoprotein (P-gp) if used systemically
* Concomitant conditions: childbearing potential without proper contraceptive measures, pregnancy, or breast feeding; hypersensitivity to investigational treatment or comparator treatment; calculated creatinine clearance (CrCl) < 30 mL/minute; hepatic disease which is associated with coagulopathy leading to a clinically relevant bleeding risk; any severe condition that would limit life expectancy to less than 6 months; planned invasive procedure with potential for uncontrolled bleeding; inability to take oral medication; ongoing drug addiction or alcohol abuse
* Any other contraindication listed in the local labeling for the comparator treatment or experimental treatment
* Participation in a study with an investigational drug or medical device within 30 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1504 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (165):
- United States (61):
  - Mobile, Alabama
  - Scottsdale, Arizona
  - East Palo Alto, California
  - El Cajon, California
  - National City, California
  - Sacramento, California
  - Santa Rosa, California
  - Torrance, California
  - New Haven, Connecticut
  - Stamford, Connecticut
  - Wilmington, Delaware
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Deltona, Florida
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Lakeland, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Orlando, Florida
  - Saint Augustine, Florida
  - Tallahassee, Florida
  - Savannah, Georgia
  - Aurora, Illinois
  - Chicago, Illinois
  - Elk Grove Village, Illinois
  - Joliet, Illinois
  - Rockford, Illinois
  - Annapolis, Maryland
  - Columbia, Maryland
  - Rockville, Maryland
  - Lincoln, Nebraska
  - North Las Vegas, Nevada
  - Bridgewater, New Jersey
  - Manalapan, New Jersey
  - Albuquerque, New Mexico
  - Buffalo, New York
  - New York, New York
  - Troy, New York
  - Asheville, North Carolina
  - Cantan, Ohio
  - Cleveland, Ohio
  - Mansfield, Ohio
  - Toledo, Ohio
  - Beaver, Pennsylvania
  - Butler, Pennsylvania
  - Doylestown, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Rapid City, South Dakota
  - Johnson City, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Sam Houston, Texas
  - Tyler, Texas
  - Layton, Utah
  - Bellingham, Washington
  - Burien, Washington
  - Wausau, Wisconsin
- Belgium (6):
  - Leuven, Vlaams Brabant
  - Bruxelles - Brussel
  - Gilly
  - Hasselt
  - Liège
  - Mol
- Brazil (4):
  - Curitiba, Paraná
  - Porto Alegre, Rio Grande do Sul
  - Campinas, São Paulo
  - São Paulo, São Paulo
- Canada (8):
  - Edmonton, Alberta
  - Victoria, British Columbia
  - Saint John, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Hamilton, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- China (10):
  - Guangzhou, Guangdong
  - Wuhan, Hubei
  - Changsha, Hunan
  - Nanchang, Jiangxi
  - Changchun, Jilin
  - Xi'an, Shaanxi
  - Ürümqi, Xinjiang
  - Beijing
  - Shanghai
  - Shenyang
- Denmark (4):
  - Hellerup
  - Herning
  - København NV
  - Viborg
- Finland (9):
  - Helsinki
  - Jyväskylä
  - Lappeenranta
  - Oulu
  - Pori
  - Rovaniemi
  - Tampere
  - Turku
  - Vaasa
- France (7):
  - Arras
  - Lille
  - Paris
  - Pessac
  - Toulouse
  - Tours
  - Vandœuvre-lès-Nancy
- Germany (11):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Nuremberg, Bavaria
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Bad Oeynhausen, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Mönchengladbach, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Dresden, Saxony
  - Leipzig, Saxony
  - Berlin, State of Berlin
- Greece (4):
  - Alexandroupoli
  - Attica / Athens
  - Heraklion
  - Thessaloniki
- Italy (8):
  - Acquaviva delle Fonti, Bari
  - San Fermo della Battaglia, Como
  - San Donato Milanese, Milano
  - Mestre, Venezia
  - Ancona
  - Catania
  - Roma
  - Torino
- Netherlands (5):
  - Arnhem
  - Haarlem
  - Heerlen
  - Leeuwarden
  - Maastricht
- Portugal (6):
  - Martinho Do Bispo, Coimbra District
  - Faro, Faro District
  - Carnaxide, Lisbon District
  - Almada
  - Lisbon
  - Vila Nova de Gaia
- Singapore, Singapore
- South Africa (7):
  - Alberton, Gauteng
  - Soweto, Gauteng
  - Cape Town, Western Cape
  - Kuils River, Western Cape
  - Somerset West, Western Cape
  - Worcester, Western Cape
  - Bloemfontein
- Spain (6):
  - Barcelona, Barcelona
  - Sabadell, Barcelona
  - Granada, Granada
  - Madrid, Madrid
  - Majadahonda, Madrid
  - Pamplona, Pamplona
- United Kingdom (8):
  - Chesterfield, Derbyshire
  - Bournemouth, Dorset
  - Welwyn Garden City, Hertfordshire
  - Leicester, Leicestershire
  - Nottingham, Nottinghamshire
  - Cliftonville
  - London
  - Portsmouth

REFERENCES:
- [Background] Cappato R, Ezekowitz MD, Klein AL, Camm AJ, Ma CS, Le Heuzey JY, Talajic M, Scanavacca M, Vardas PE, Kirchhof P, Hemmrich M, Lanius V, Meng IL, Wildgoose P, van Eickels M, Hohnloser SH; X-VeRT Investigators. Rivaroxaban vs. vitamin K antagonists for cardioversion in atrial fibrillation. Eur Heart J. 2014 Dec 14;35(47):3346-55. doi: 10.1093/eurheartj/ehu367. Epub 2014 Sep 2. PMID 25182247
- [Background] Hai Z, Guangrui S. Cardiac paraganglioma. Eur Heart J. 2018 Jun 14;39(23):2219. doi: 10.1093/eurheartj/ehu241. No abstract available. PMID 24944325
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 141 centers (involving 144 investigators) in Europe, South Africa, North America, and Asia Pacific.
Pre-assignment Details: Overall, 1584 subjects were screened and 80 subjects did not complete or pass screening. 1504 subjects were randomized; 1002 were assigned to rivaroxaban and 502 to vitamin K antagonist (VKA).
Groups:
- Rivaroxaban (Xarelto, BAY59-7939): Subjects randomized to treatment with rivaroxaban received rivaroxaban 20 milligram (mg) orally once daily. Subjects with moderate renal impairment [i.e., Creatinine clearance (CrCl) of 30 to 49 milliliter per minute (mL/min), inclusive] at screening received the adjusted dose of 15 mg once daily. The duration of the treatment period for a given subject depended on the cardioversion strategy. For subjects in the Direct Cardioversion Strategy, the cardioversion procedure was performed within 1-5 days after randomization. Rivaroxaban was given for 1-5 days before planned direct cardioversion and for 42 days thereafter. Subjects in the Delayed Cardioversion Strategy received rivaroxaban for 21 (+4) to 56 (+4) days prior to cardioversion and for 42 days thereafter. The investigator assessed whether or not long-term anticoagulation was warranted and treated the subject according to standard of care. Then subjects entered 30-day follow-up period.
- Vitamin K Antagonist (VKA): Subjects assigned to treatment with VKA received VKA orally once daily titrated to a target INR of 2.5 (range 2.0-3.0, inclusive). The specific VKA was given by the investigator based on local standard of practice. For all subjects randomized to receive VKA, the investigator assessed if a parenteral anticoagulant drug, particularly before cardioversion, was needed as bridging therapy with VKA as standard of care (until target INR was achieved). The duration depended on the cardioversion strategy. For subjects in the Direct Cardioversion Strategy, cardioversion was performed within 1-5 days after randomization. VKA was given for 1-5 days before it and for 42 days thereafter. Subjects in the Delayed Cardioversion Strategy received VKA for 21 (+4) to 56 (+4) days before cardioversion and for 42 days thereafter. The investigator assessed if long-term anticoagulation was warranted and treated the subject according to standard of care or not. Then subjects entered 30-day follow-up period.
Period: Treatment Period
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Vitamin K Antagonist (VKA)
Started | 1002 | 502
Subjects Received Treatment | 988 | 499
Completed | 846 | 400
Not Completed | 156 | 102
Not completed — Death | 4 | 1
Not completed — Efficacy outcome reached | 0 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Adverse Event | 60 | 22
Not completed — Non-compliance with study drug | 3 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 19 | 16
Not completed — Switching to other therapy | 5 | 2
Not completed — Logistical difficulties | 5 | 8
Not completed — Treatment failure | 0 | 14
Not completed — Protocol Violation | 56 | 36
Period: 30-day Safety Follow-up Period
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Vitamin K Antagonist (VKA)
Started | 982 | 487
Completed | 924 | 446
Not Completed | 58 | 41
Not completed — Death | 3 | 2
Not completed — Non-compliance with study drug | 0 | 1
Not completed — Protocol Violation | 39 | 22
Not completed — Logistical difficulties | 1 | 3
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Lost to Follow-up | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Vitamin K Antagonist (VKA) | Total
Number analyzed (Participants) | 1002 | 502 | 1504
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (10.6) | 64.7 (10.5) | 64.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 135 | 410
  Male | 727 | 367 | 1094
CHADS 2 score [Mean (Standard Deviation); unit: units on scale] — Predicts clinical risk of stroke and thromboembolism in atrial fibrillation incorporating these risk factors: Congestive heart failure, Hypertension, Age [greater than or equal to (>=)75 years], Diabetes mellitus, Stroke/transient ischemic attack. Total score ranged from 0 to 6, with "0"= low risk, "1"= moderate risk and ">=2"= high risk.
  units on scale | 1.3 (1.1) | 1.4 (1.1) | 1.4 (1.1)
CHA 2 DS 2 VASc score [Mean (Standard Deviation); unit: units on scale] — Predicts clinical risk of stroke and thromboembolism in atrial fibrillation incorporating these risk factors: Congestive heart failure/left ventricular dysfunction, Hypertension, Age >= 75 years, Diabetes mellitus, Stroke/transient ischemic attack/thromboembolism, Vascular disease (prior myocardial infarction, peripheral artery disease, or aortic plaque), Age 65 - 74 years, Sex category (i.e., female). Total score ranged from 0 to 8, with "0" (or 1 if female only)= Low risk ; "1" (except for female gender alone)= moderate risk and ">=2"=high risk.
  units on scale | 2.3 (1.6) | 2.3 (1.6) | 2.3 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite of the Following Events, Adjudicated Centrally: Stroke, Transient Ischemic Attack, Non-central Nervous System Systemic Embolism, Myocardial Infarction and Cardiovascular Death
Description: Stroke, TIA, Non-CNS Embolism, MI and cardiovascular death were adjudicated and confirmed by Clinical Endpoints Committee (CEC). Stroke included hemorrhagic and ischemic infarction. TIA including information if with or without matching lesion. Non CNS systemic embolism included emboli in peripheral arterial of the upper and lower extremities, ocular and retinal (pulmonary embolism and MI were excluded from the category). MI was assessed based on either cardiac biomarkers, new abnormal Q waves appeared on electrocardiogram for >= 2 leads, or autopsy confirmation. Cardiovascular death included death in subjects with non-valvular atrial fibrillation (AF). Number of subjects with composite events were reported.
Time Frame: From randomization to the date of last dose of study drug +2 days for subjects who completed planned treatment or the earlier date [last planned dose, follow-up visit at the end of 30-day follow-up period] for subjects who prematurely stopped treatment
Population: The primary population for the efficacy analysis was the modified intention-to-treat (mITT) population. mITT population included all the randomized subjects in whom a left atrial/left atrial appendage (LA/LAA) thrombus was not diagnosed during a transesophageal echocardiogram (TEE) performed before the first planned cardioversion in the study.
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 978 | 492
Participants | 5 | 5
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Vitamin K Antagonist (VKA); Descriptive comparison of crude estimates of the cumulative incidence and estimation of risk ratio, all with 95% confidence intervals; Test type: Superiority or Other; no statistical test performed; Risk Ratio (RR) = 0.50, 95% CI 2-sided [0.15 to 1.73] — Crude estimate of the cumulative incidence for rivaroxaban (Xarelto, BAY59-7939): 0.51% (0.20% - 1.17%). Crude estimate of the cumulative incidence for Vitamin K antagonist (VKA): 1.02% (0.40% - 2.34%)

2. Primary Outcome: Number of Participants With Major Bleedings as Per Central Adjudication
Description: Bleeding events were adjudicated and confirmed by CEC blinded to treatment. The CEC categorized the bleeding events as major or non-major. The bleeding events were defined per the International Society on Thrombosis and Hemostasis (ISTH) criteria. Major bleeding was clinically overt bleeding associated with a fall in hemoglobin of 2 gram per deciliter (g/dL) or higher, leading to a transfusion of 2 or more units of packed red blood cells or whole blood, occurring in a critical site or contributing to death. Number of subjects with confirmed adjudicated bleeding events occurring in greater than (>)1 total subjects were reported.
Time Frame: From randomization up to the date of the last dose of study drug + 2 days
Population: The safety profile was analyzed using the safety analysis set (SAF) population. SAF population included all randomized subjects who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 988 | 499
Participants | 6 | 4
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Vitamin K Antagonist (VKA); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; no test performed; Risk Ratio (RR) = 0.76, 95% CI 2-sided [0.21 to 2.67] — Crude estimate of the cumulative incidence for rivaroxaban (Xarelto, BAY59-7939): 0.61% (0.26% - 1.27%). Crude estimate of the cumulative incidence for Vitamin K antagonist (VKA): 0.80% (0.27% - 2.00%)

3. Secondary Outcome: Number of Participants With Composite of Strokes and Non-central Nervous System Systemic Embolisms
Description: Stroke and Non-CNS Embolism were adjudicated and confirmed by CEC. Stroke included hemorrhagic and ischemic infarction. Non CNS systemic embolism included emboli in peripheral arterial of the upper and lower extremities, ocular and retinal (pulmonary embolism and MI were excluded from the category). Number of subjects with composite events were reported.
Time Frame: as for outcome 1
Population: The primary population for the efficacy analysis was the mITT population. mITT population included all the randomized subjects in whom a LA/LAA thrombus was not diagnosed during a TEE performed before the first planned cardioversion in the study.
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 978 | 492
Participants | 2 | 3
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Vitamin K Antagonist (VKA); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; no statistical test performed; Risk Ratio (RR) = 0.34, 95% CI 2-sided [0.06 to 2.00] — Crude estimate of the cumulative incidence for rivaroxaban (Xarelto, BAY59-7939): 0.20% (0.04% - 0.71%). Crude estimate of the cumulative incidence for Vitamin K antagonist (VKA): 0.61% (0.17% - 1.72%)

4. Secondary Outcome: Number of Participants With Composite of Strokes, Transient Ischemic Attacks, Non-central Nervous System Systemic Embolisms, Myocardial Infarctions and All-cause Mortality
Description: Stroke, TIA, Non- CNS systemic embolism, MI and all-cause mortality were adjudicated and confirmed by CEC. Stroke included hemorrhagic and ischemic infarction. TIA including information if with or without matching lesion. Non CNS systemic embolism included emboli in peripheral arterial of the upper and lower extremities, ocular and retinal (pulmonary embolism and MI were excluded from the category). MI was assessed based on either cardiac biomarkers, new abnormal Q waves appeared on electrocardiogram for >= 2 leads, or autopsy confirmation. All-cause mortality included vascular death and non-vascular death. Number of subjects with composite events were reported.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 978 | 492
Participants | 6 | 6
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Vitamin K Antagonist (VKA); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; no statistical test performed; Risk Ratio (RR) = 0.50, 95% CI 2-sided [0.16 to 1.55] — Crude estimate of the cumulative incidence for rivaroxaban (Xarelto, BAY59-7939): 0.61% (0.27% - 1.29%). Crude estimate of the cumulative incidence for Vitamin K antagonist (VKA): 1.22% (0.53% - 2.51%)

5. Secondary Outcome: Number of Participants With Strokes
Description: All events were adjudicated and confirmed by a CEC blinded to treatment. Stroke included hemorrhagic (Stroke with local collections of intraparenchymal blood. Subarachnoid hemorrhage, subdural hemorrhage, and epidural hemorrhage were excluded), ischemic infarction (Stroke without focal collection of intracranial blood) and unknown (No imaging data and anatomic findings were available). Number of subjects with strokes were reported.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 978 | 492
Participants | 2 | 2

6. Secondary Outcome: Number of Participants With Transient Ischemic Attacks
Description: All events were adjudicated and confirmed by a CEC blinded to treatment. Number of subjects with TIA were reported.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 978 | 492
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Non-central Nervous System Systemic Embolisms
Description: All events were adjudicated and confirmed by a CEC blinded to treatment. Non CNS systemic embolism included emboli in peripheral arterial of the upper and lower extremities, ocular and retinal (pulmonary embolism and MI were excluded from the category). Number of subjects with non-CNS embolism were reported.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 978 | 492
Participants | 0 | 1

8. Secondary Outcome: Number of Participants With Myocardial Infarctions
Description: All events were adjudicated and confirmed by a CEC blinded to treatment. MI was assessed based onmeither cardiac biomarkers, new abnormal Q waves appeared on electrocardiogram for >= 2 leads, or autopsy confirmation. Number of subjects with MI were reported.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 978 | 492
Participants | 1 | 1

9. Secondary Outcome: Number of Participants With Cardiovascular Deaths
Description: All events were adjudicated and confirmed by a CEC blinded to treatment. Any death that was not clearly non-vascular (e.g., deaths due to spontaneous bleeding, myocardial infarction, stroke, cardiac failure, and arrhythmia). Number of subjects with cardiovascular deaths were reported.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 978 | 492
Participants | 4 | 2
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Vitamin K Antagonist (VKA); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; no statistical test performed; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.18 to 5.47] — Crude estimate of the cumulative incidence for rivaroxaban (Xarelto, BAY59-7939): 0.41% (0.14% - 1.02%). Crude estimate of the cumulative incidence for Vitamin K antagonist (VKA): 0.41% (0.07% - 1.41%)

10. Secondary Outcome: Number of Participants With All-cause Mortality
Description: All events were adjudicated and confirmed by a CEC blinded to treatment. All-cause mortality included vascular death and non-vascular death. Number of subjects with all-cause mortality were reported.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 978 | 492
Participants | 5 | 3
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Vitamin K Antagonist (VKA); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; no statistical test performed; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.20 to 3.49] — Crude estimate of the cumulative incidence for rivaroxaban (Xarelto, BAY59-7939): 0.51% (0.20% - 1.17%). Crude estimate of the cumulative incidence for Vitamin K antagonist (VKA): 0.61% (0.17% - 1.72%)

11. Secondary Outcome: Number of Participants With Composite of Major and Non-major Bleeding Events
Description: All events were adjudicated and confirmed by a CEC blinded to treatment. The CEC categorized the bleeding events as major or non-major. The bleeding events were defined per the ISTH criteria. Clinically relevant bleeding included major bleeding (overt bleeding associated with 2 g/dL or greater fall in hemoglobin, leading to a transfusion of 2 or more units of packed red blood cells or whole blood, occurring in a critical site or contributing to death) and non-major bleeding associated with medical intervention, unscheduled physician contact, (temporary) cessation of study treatment, discomfort for the participants such as pain, or impairment of activities of daily life. Number of subjects with clinically relevant major and non-major bleeding events were reported.
Time Frame: From randomization up to the date of the last dose of study drug + 2 days
Population: The safety profile was analyzed using the SAF population. SAF population included all randomized subjects who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 988 | 499
Participants | 33 | 14

ADVERSE EVENTS:
Time Frame: From first administration of study drug to date of last study drug + 2 days
Groups:
- Rivaroxaban (Xarelto; BAY59-7939): Subjects randomized to treatment with rivaroxaban received rivaroxaban 20 milligram (mg) orally once daily. Subjects with moderate renal impairment [i.e., Creatinine clearance (CrCl) of 30 to 49 milliliter per minute (mL/min), inclusive] at screening received the adjusted dose of 15 mg once daily. The duration of the treatment period for a given subject depended on the cardioversion strategy. For subjects in the Direct Cardioversion Strategy, the cardioversion procedure was performed within 1-5 days after randomization. Rivaroxaban was given for 1-5 days before planned direct cardioversion and for 42 days thereafter. Subjects in the Delayed Cardioversion Strategy received rivaroxaban for 21 (+4) to 56 (+4) days prior to cardioversion and for 42 days thereafter. The investigator assessed whether or not long-term anticoagulation was warranted and treated the subject according to standard of care. Then subjects entered 30-day follow-up period.
- Vitamin K Antagonist: Subjects assigned to treatment with VKA received VKA orally once daily titrated to a target INR of 2.5 (range 2.0-3.0, inclusive). The specific VKA was given by the investigator based on local standard of practice. For all subjects randomized to receive VKA, the investigator assessed if a parenteral anticoagulant drug, particularly before cardioversion, was needed as bridging therapy with VKA as standard of care (until target INR was achieved). The duration depended on the cardioversion strategy. For subjects in the Direct Cardioversion Strategy, cardioversion was performed within 1-5 days after randomization. VKA was given for 1-5 days before it and for 42 days thereafter. Subjects in the Delayed Cardioversion Strategy received VKA for 21 (+4) to 56 (+4) days before cardioversion and for 42 days thereafter. The investigator assessed if long-term anticoagulation was warranted and treated the subject according to standard of care or not. Then subjects entered 30-day follow-up period.
Arm/Group | Rivaroxaban (Xarelto; BAY59-7939) | Vitamin K Antagonist
Serious Adverse Events (participants affected / at risk) | 93/988 | 38/499
Other Adverse Events (participants affected / at risk) | 272/988 | 126/499
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (Xarelto; BAY59-7939) (N=988) | Vitamin K Antagonist (N=499)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 8 | 4
Atrial flutter (Cardiac disorders) | 4 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 4 | 3
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 3 | 3
Cardiac arrest (Cardiac disorders) | 3 | 0
Cardiac failure (Cardiac disorders) | 8 | 2
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 10 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 3 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Rhythm idioventricular (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 2
Tachycardia induced cardiomyopathy (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Blindness transient (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 5 | 0
Medical device site reaction (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Bronchitis viral (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 3
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arteriogram coronary (Investigations) | 0 | 1
Electrocardiogram PR prolongation (Investigations) | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Thalamus haemorrhage (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 2
Urogenital haemorrhage (Renal and urinary disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bladder catheterisation (Surgical and medical procedures) | 0 | 1
Cardiac ablation (Surgical and medical procedures) | 3 | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 1 | 0
Plastic surgery (Surgical and medical procedures) | 0 | 1
Shoulder arthroplasty (Surgical and medical procedures) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (Xarelto; BAY59-7939) (N=988) | Vitamin K Antagonist (N=499)
Atrial fibrillation (Cardiac disorders) | 2 | 7
Atrial thrombosis (Cardiac disorders) | 16 | 6
Atrioventricular block first degree (Cardiac disorders) | 40 | 25
Bradycardia (Cardiac disorders) | 30 | 13
Sinus bradycardia (Cardiac disorders) | 25 | 12
Constipation (Gastrointestinal disorders) | 10 | 3
Diarrhoea (Gastrointestinal disorders) | 18 | 3
Nausea (Gastrointestinal disorders) | 17 | 1
Fatigue (General disorders) | 14 | 9
Oedema peripheral (General disorders) | 20 | 5
Influenza (Infections and infestations) | 3 | 5
Nasopharyngitis (Infections and infestations) | 12 | 5
Urinary tract infection (Infections and infestations) | 7 | 5
Contusion (Injury, poisoning and procedural complications) | 3 | 5
International normalised ratio increased (Investigations) | 1 | 9
Dizziness (Nervous system disorders) | 25 | 9
Headache (Nervous system disorders) | 25 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 30 | 9
Rash (Skin and subcutaneous tissue disorders) | 12 | 5
Hypertension (Vascular disorders) | 22 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Consultant agrees not to publish or cause to be published any works of authorship relating to the Project rendered pursuant to this Agreement without first notifying Bayer in writing and obtaining Bayer's written consent. Bayer will respond to such notification within sixty (60) days of receipt.Bayer reserves the right to insist on the removal of all or any of its Confidential Information from any such work prior to publication